CLINICAL TRIAL: NCT02713997
Title: Anti-inflammatory Therapy to Improve Outcomes in Patients With Chronic Pancreatitis Undergoing Total Pancreatectomy Islet Autotransplantation
Brief Title: Anti-inflammatory Therapy to Improve Outcomes After TPIAT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PEDS-2016-22934; R01DK109914 (NIH)
Record Dates: First submitted 2016-02-29; First posted 2016-03-21 (Estimated); Results first posted 2024-09-26 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Pancreatitis, Chronic; Diabetes; Transplant
MeSH Terms: conditions — Pancreatitis; Bronchiolitis Obliterans Syndrome; Diabetes Mellitus | interventions — Etanercept; alpha 1-Antitrypsin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Standard Care (No Intervention): Patients in the standard care arm will undergo the usual procedure of TPIAT with no ancillary therapies provided.
- etanercept (Experimental): Patients in the etanercept arm will undergo the usual procedure of TPIAT with additional therapy of etanercept.
  Interventions: Drug: etanercept
- alpha-1 antitrypsin (Experimental): Patients in the alpha-1 antitrypsin arm will undergo the usual procedure of TPIAT with additional therapy of alpha-1 antitrypsin (Aralast NP)
  Interventions: Drug: Alpha 1-Antitrypsin

INTERVENTIONS:
Drug: etanercept — 50 mg on day 0 SQ; 25 mg subcutaneous (SQ) on days 3, 7, 10, 14, and 21 relative to TPIAT
  Other Names: Enbrel
  Arms: etanercept
Drug: Alpha 1-Antitrypsin — 90 mg/kg intravenous infusion on days -1, and +3, 7, 14, 21, and 28 post-transplant
  Other Names: Aralast NP
  Arms: alpha-1 antitrypsin

SUMMARY:
Patients with severe chronic pancreatitis may be candidates to have their pancreas removed and their islets transplanted into the liver to reduce the risk of diabetes mellitus, a procedure called total pancreatectomy with islet autotransplant (TPIAT). However, over half of patients who have a TPIAT will need to remain on some supplemental insulin life-long after the procedure. We will study therapies that may reduce damage to transplanted islets, and thereby improve long-term outcomes.

Two promising anti-inflammatory therapies are available to protect islets from damage at the time of transplant: (1) the Tumor Necrosis Factor (TNF)-alpha inhibitor etanercept and (2) the serine protease inhibitor alpha-1 antitrypsin. Both agents are commercially available for clinical trials. Proof-of-principle for etanercept has been demonstrated in type 1 diabetic allotransplant recipients, in whom a 10 day course of etanercept early post-transplant significantly improved long-term insulin independence, due to better survival of the transplanted beta cell mass in the engraftment period. Alpha-1 antitrypsin (A1AT) reduces inflammatory cytokines, protects against cytokine-induced beta cell apoptosis, and prolongs islet graft survival in mice and intraportal IAT non-human primates.

This initial 3-arm drug-treatment clinical trial will investigate the use of Etanercept and A1AT to improve IAT function at 90 days and 1 and 2 years post-TPIAT compared to standard care. Forty-five patients undergoing TPIAT will be randomized 1:1:1 to receive either: 1) etanercept (50 mg on day 0; 25 mg on days 3, 7, 10, 14, and 21), 2) alpha-1 antitrypsin (90 mg/kg IV days -1, +3, 7, 14, 21, 28) or 3) standard care. Patients will have mechanistic assessments drawn in the early post-operative period including inflammatory cytokines and chemokines and measures of beta cell loss. Metabolic testing will occur at 90, 365, and 730 days post-TPIAT, including mixed meal tolerance testing, IV glucose tolerance testing, and glucose-potentiated arginine-induced insulin secretion (GPAIS).

DETAILED DESCRIPTION:
For patients with severe pancreatitis refractory to medical and endoscopic therapy, total pancreatectomy (TP) with islet autotransplantation (IAT) may be considered. While 90% of TPIAT recipients have some function of the transplanted islet graft, only about 1/3rd come completely off insulin. The long-term goal of the proposed research is to develop new therapies that will increase the number of patients who are non-diabetic following islet autotransplant. Such therapies may also benefit recipients of islet allotransplant for type 1 diabetes.

Following islet transplantation, the islets must acutely survive the stress of the procedure, and then they must engraft in the liver and establish a vascular supply. The greater the functional islet mass engrafted, the lower the risk of post-operative diabetes. It has been estimated that more than half of the islet mass may be lost in the early post-transplant period in islet transplant recipients. Beta cell apoptosis is common during the first month post-transplant and is upregulated in the presence of inflammatory cytokines such as TNF-alpha. Thus, a major contributor to islet loss is the inflammatory damage sustained by the transplanted islets in the early post-transplant period; we propose to directly target this destructive process.

Two promising anti-inflammatory therapies are available to address this problem: (1) the TNF-alpha inhibitor etanercept and (2) the serine protease inhibitor alpha-1 antitrypsin. Both agents are commercially available for clinical trials. Proof-of-principle for etanercept has been demonstrated in type 1 diabetic allotransplant recipients, in whom a 10 day course of etanercept early post-transplant significantly improved long-term insulin independence, due to better survival of the transplanted beta cell mass in the engraftment period. Alpha-1 antitrypsin (A1AT) reduces inflammatory cytokines, protects against cytokine-induced beta cell apoptosis, and prolongs islet graft survival in mice and intraportal IAT non-human primates.

This initial 3-arm drug-treatment clinical trial will investigate the use of Etanercept and A1AT to improve IAT function at 90 days and 1 and 2 years post-TPIAT compared to standard care. Forty-five patients undergoing TPIAT will be randomized 1:1:1 to receive either: 1) etanercept (50 mg on day 0; 25 mg on days 3, 7, 10, 14, and 21), 2) alpha-1 antitrypsin (90 mg/kg IV days -1, +3, 7, 14, 21, 28) or 3) standard care. Patients will have mechanistic assessments drawn in the early post-operative period including inflammatory cytokines and chemokines and measures of beta cell loss. Metabolic testing will occur at 90, 365, and 730 days post-TPIAT, including mixed meal tolerance testing, IV glucose tolerance testing, and glucose-potentiated arginine-induced insulin secretion (GPAIS). The latter measures the maximally stimulated acute C-peptide response (ACRmax) as the best estimate of islet mass and the primary endpoint (at day 90) for this study. Results will be used to select the most promising agent for future study in a randomized, blinded multi-center clinical trial.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18- 68 years. .
2. Scheduled for total pancreatectomy and IAT at University of Minnesota (UM). All patients who are approved for pancreatectomy and IAT at UM are reviewed by a multi-disciplinary committee including surgeons, gastroenterologists specializing in pancreatic disease, a pain specialist, psychologist, and endocrinologist to confirm the diagnosis of chronic pancreatitis and candidate suitability for surgery.
3. Able to provide informed consent

Exclusion Criteria:

1. Pre-existing diagnosis of diabetes mellitus, fasting blood glucose >115 mg/dl, or hemoglobin A1c level >6.0% because these are all evidence of inadequate beta-cell mass.
2. Use of any of the following treatments in the 30 days prior to enrollment: insulin, metformin, sulfonylureas, glinides, thiazolidinediones, Glucagon Like Peptide (GLP)-1 agonists, dipeptidyl peptidase (DPP-4) inhibitors, or amylin.
3. Immunoglobulin (IgA) deficiency (serum level <5 mg/dL), which has been associated with hypersensitivity to alpha-1 antitrypsin.
4. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST)>2.5 times the upper limit of normal (ULN). Bilirubin >ULN, unless due to benign diagnosis such as Gilbert's.
5. Known history of human immunodeficiency virus (HIV) infection, hepatitis B (chronic), or hepatitis C (chronic).
6. History of tuberculosis (TB) (latent or active disease), or positive TB skin test.
7. History of symptomatic fungal lung infection.
8. History of multiple sclerosis, transverse myelitis, Guillain Barre, or other suspected demyelinating disease, due to risk of exacerbation of these conditions with use of etanercept; or prior history of systemic lupus erythematosus
9. Any of the following hematologic abnormalities: severe anemia (hgb <10 g/dL), thrombocytopenia (<150/mm3), or neutropenia (<1.0 x109/L).
10. Current use or expected use of oral or injected corticosteroids, or any mediation likely to affect glucose tolerance. However, use of hydrocortisone for physiologic replacement, or use of any topical, inhaled, or intranasal glucocorticoid is permitted.
11. Current or expected use of any other immunosuppressive agent.
12. Known hypersensitivity to etanercept or A1AT.
13. Any condition that is likely, in the opinion of the patient's medical providers, to necessitate use of TNF alpha therapeutically in the future (such as psoriatic arthritis).
14. Known coagulopathy, or need for anticoagulant therapy preoperatively (coumadin, enoxaparin), or any history of pulmonary embolism.
15. For females, plans to become pregnant or unwillingness to use birth control for the study duration.
16. Inability to comply with the study protocol.
17. Untreated psychiatric illness that may interfere with ability to give informed consent, or other developmental delay or neurocognitive disorder that impairs with a patient's ability to consent on their own behalf.
18. Any other medical condition that, in the opinion of the investigator, may interfere with the patient's ability to successfully and safely complete the trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2025-05-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard Care | Etanercept | Alpha-1 Antitrypsin
Started | 16 | 14 | 13
Completed | 16 | 14 | 13
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Care | Etanercept | Alpha-1 Antitrypsin | Total
Number analyzed (Participants) | 16 | 14 | 13 | 43
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 16 | 14 | 13 | 43
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.4 (12.1) | 40.8 (12) | 37.3 (12.6) | 38.5 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 10 | 3 | 26
  Male | 3 | 4 | 10 | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 1
  White | 16 | 11 | 13 | 40
  More than one race | 0 | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Maximal Acute C-peptide Response to Glucose (ACRmax)
Description: derived from times 0-5 minute C-peptide measures on glucose potentiated arginine stimulation at day 90 post-TPIAT
Time Frame: day 90
Measure: Mean (Standard Deviation); unit: ng/mL*min
Arm/Group | Standard Care | Etanercept | Alpha-1 Antitrypsin
Number analyzed (Participants) | 15 | 14 | 13
ng/mL*min | 1.06 (0.26) | 1.52 (0.28) | 1.29 (0.28)

2. Secondary Outcome: ACRmax
Description: derived from times 0- 5 minute C-peptide values from glucose potentiated arginine
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: ng/mL*min
Arm/Group | Standard Care | Etanercept | Alpha-1 Antitrypsin
Number analyzed (Participants) | 15 | 14 | 11
ng/mL*min | 1.16 (0.32) | 1.44 (0.33) | 1.88 (0.39)

3. Secondary Outcome: Maximal Acute Insulin Response to Glucose (AIRmax)
Description: derived from times 0- 5 minute insulin values from glucose potentiated arginine
Time Frame: day 90
Measure: Mean (Standard Deviation); unit: mU/L*min
Arm/Group | Standard Care | Etanercept | Alpha-1 Antitrypsin
Number analyzed (Participants) | 15 | 14 | 13
mU/L*min | 24.85 (6.26) | 34.96 (6.99) | 30.43 (6.72)

4. Secondary Outcome: Insulin Independence
Description: no insulin use for >14 days
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Care | Etanercept | Alpha-1 Antitrypsin
Number analyzed (Participants) | 16 | 14 | 13
Participants | 2 | 4 | 2

5. Secondary Outcome: Insulin Dose (Unit/Day)
Description: calculated by average daily insulin dose from 2 weeks of logs
Time Frame: day 90
Measure: Mean (Standard Deviation); unit: unit/day
Arm/Group | Standard Care | Etanercept | Alpha-1 Antitrypsin
Number analyzed (Participants) | 15 | 14 | 13
unit/day | 22.3 (4.3) | 17.2 (4.6) | 26 (4.7)

6. Secondary Outcome: Area Under the Curve (AUC) C-peptide
Description: calculated as area under the curve from every 30 minute C-peptide values on mixed meal tolerance test (MMTT)
Time Frame: day 90, 1 year, 2 years
Reporting Status: Not Posted

7. Secondary Outcome: AUC Glucose
Description: calculated as area under the curve from every 30 minute glucose values on MMTT
Time Frame: day 90, 1 year, 2 years
Reporting Status: Not Posted

8. Secondary Outcome: Absence of Severe Hypoglycemia (SHE) With A1c <7%
Description: no events meeting American Diabetes Association (ADA criteria for SHE day 28- 365, and day 365- 730 respectively with A1c value of <7%
Time Frame: 1 year, 2 years
Reporting Status: Not Posted

9. Secondary Outcome: Severe Adverse Events
Time Frame: cumulative, through 2 year visit
Reporting Status: Not Posted

10. Secondary Outcome: ACRmax
Description: derived from times 0- 5 minute C-peptide values from glucose potentiated arginine
Time Frame: 2 year
Measure: Mean (Standard Deviation); unit: ng/mL*min
Arm/Group | Standard Care | Etanercept | Alpha-1 Antitrypsin
Number analyzed (Participants) | 13 | 10 | 8
ng/mL*min | 1.38 (0.45) | 2.03 (0.51) | 2.6 (0.57)

11. Secondary Outcome: Maximal Acute Insulin Response to Glucose (AIRmax)
Description: derived from times 0- 5 minute insulin values from glucose potentiated arginine
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: mU/L*min
Arm/Group | Standard Care | Etanercept | Alpha-1 Antitrypsin
Number analyzed (Participants) | 15 | 14 | 11
mU/L*min | 28.4 (9) | 37.2 (9.4) | 44.6 (11)

12. Secondary Outcome: Maximal Acute Insulin Response to Glucose (AIRmax)
Description: derived from times 0- 5 minute insulin values from glucose potentiated arginine
Time Frame: 2 year
Measure: Mean (Standard Deviation); unit: mU/L*min
Arm/Group | Standard Care | Etanercept | Alpha-1 Antitrypsin
Number analyzed (Participants) | 13 | 10 | 8
mU/L*min | 34.3 (11.8) | 47.4 (13.5) | 56.9 (15.1)

13. Secondary Outcome: Insulin Independence
Description: no insulin use for >14 days
Time Frame: 2 year
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Care | Etanercept | Alpha-1 Antitrypsin
Number analyzed (Participants) | 16 | 14 | 12
Participants | 2 | 5 | 2

14. Secondary Outcome: Insulin Dose (Unit/Day)
Description: calculated by average daily insulin dose from 2 weeks of logs
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: unit/day
Arm/Group | Standard Care | Etanercept | Alpha-1 Antitrypsin
Number analyzed (Participants) | 15 | 14 | 13
unit/day | 15.7 (3.8) | 12 (4) | 24.4 (4.4)

15. Secondary Outcome: Insulin Dose (Unit/Day)
Description: calculated by average daily insulin dose from 2 weeks of logs
Time Frame: 2 year
Measure: Mean (Standard Deviation); unit: unit/day
Arm/Group | Standard Care | Etanercept | Alpha-1 Antitrypsin
Number analyzed (Participants) | 15 | 14 | 11
unit/day | 13 (3.5) | 16.8 (3.9) | 16.1 (4.3)

16. Secondary Outcome: Area Under the Curve (AUC) C-peptide
Description: calculated as area under the curve from every 30 minute C-peptide values on mixed meal tolerance test (MMTT)
Time Frame: 90 days
Measure: Mean (Standard Deviation); unit: ng/mL*min
Arm/Group | Standard Care | Etanercept | Alpha-1 Antitrypsin
Number analyzed (Participants) | 15 | 14 | 13
ng/mL*min | 186.6 (29.44) | 247.6 (30.47) | 171.9 (31.6)

17. Secondary Outcome: Area Under the Curve (AUC) C-peptide
Description: calculated as area under the curve from every 30 minute C-peptide values on mixed meal tolerance test (MMTT)
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: ng/mL*min
Arm/Group | Standard Care | Etanercept | Alpha-1 Antitrypsin
Number analyzed (Participants) | 15 | 14 | 11
ng/mL*min | 192 (39) | 257 (40) | 223 (45)

18. Secondary Outcome: Area Under the Curve (AUC) C-peptide
Description: calculated as area under the curve from every 30 minute C-peptide values on mixed meal tolerance test (MMTT)
Time Frame: 2 year
Measure: Mean (Standard Deviation); unit: ng/mL*min
Arm/Group | Standard Care | Etanercept | Alpha-1 Antitrypsin
Number analyzed (Participants) | 13 | 10 | 9
ng/mL*min | 165 (39) | 276 (44) | 235 (47)

19. Secondary Outcome: AUC Glucose
Description: calculated as area under the curve from every 30 minute glucose values on MMTT
Time Frame: 90 days
Measure: Mean (Standard Error); unit: mg/dL*min
Arm/Group | Standard Care | Etanercept | Alpha-1 Antitrypsin
Number analyzed (Participants) | 15 | 14 | 13
mg/dL*min | 18404 (1245) | 18144 (1289) | 19734 (1338)

20. Secondary Outcome: AUC Glucose
Description: calculated as area under the curve from every 30 minute glucose values on MMTT
Time Frame: 1 year
Measure: Mean (Standard Error); unit: mg/dL*min
Arm/Group | Standard Care | Etanercept | Alpha-1 Antitrypsin
Number analyzed (Participants) | 15 | 14 | 11
mg/dL*min | 21099 (1558) | 20770 (1612) | 21712 (1819)

21. Secondary Outcome: AUC Glucose
Description: calculated as area under the curve from every 30 minute glucose values on MMTT
Time Frame: 2 year
Measure: Mean (Standard Error); unit: mg/dL*min
Arm/Group | Standard Care | Etanercept | Alpha-1 Antitrypsin
Number analyzed (Participants) | 13 | 10 | 9
mg/dL*min | 21493 (1921) | 18040 (2190) | 21846 (2309)

22. Secondary Outcome: Absence of Severe Hypoglycemia (SHE) With A1c <7%
Description: no events meeting American Diabetes Association (ADA criteria for SHE day 28- 365)
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Care | Etanercept | Alpha-1 Antitrypsin
Number analyzed (Participants) | 15 | 14 | 11
Participants | 11 | 10 | 10

23. Secondary Outcome: Absence of Severe Hypoglycemia (SHE) With A1c <7%
Description: no events meeting American Diabetes Association (ADA criteria for SHE day 28- 365)
Time Frame: 2 year
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Care | Etanercept | Alpha-1 Antitrypsin
Number analyzed (Participants) | 13 | 13 | 11
Participants | 9 | 9 | 6

ADVERSE EVENTS:
Time Frame: collected over 90 days for all AE and 1 year for SAE
Arm/Group | Standard Care | Etanercept | Alpha-1 Antitrypsin
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/14 | 0/13
Serious Adverse Events (participants affected / at risk) | 12/16 | 4/14 | 4/13
Other Adverse Events (participants affected / at risk) | 14/16 | 13/14 | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Care (N=16) | Etanercept (N=14) | Alpha-1 Antitrypsin (N=13)
abdominal infection (General disorders) | 0 (0) | 1 (1) | 1 (2)
abdominal pain (General disorders) | 2 (3) | 2 (10) | 4 (4)
diarrhea (General disorders) | 1 (1) | 2 (3) | 0 (0)
ALT/AST elevated (General disorders) | 1 (1) | 0 (0) | 0 (0)
fever (General disorders) | 2 (2) | 1 (1) | 0 (0)
heme: clot or bleed (General disorders) | 1 (1) | 2 (3) | 0 (0)
hypotension (General disorders) | 1 (1) | 0 (0) | 0 (0)
kidney/bladder issue (General disorders) | 0 (0) | 1 (1) | 0 (0)
metabolic and electrolyte abnormalities (General disorders) | 2 (2) | 0 (0) | 2 (2)
MSK pain (General disorders) | 0 (0) | 2 (2) | 0 (0)
Nausea/Vomiting (General disorders) | 1 (1) | 0 (0) | 1 (1)
other GI (General disorders) | 3 (4) | 2 (4) | 3 (3)
other infection (General disorders) | 4 (5) | 4 (7) | 4 (5)
respiratory disease (General disorders) | 0 (0) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Care (N=16) | Etanercept (N=14) | Alpha-1 Antitrypsin (N=13)
abdominal infection (General disorders) | 1 (1) | 1 (1) | 1 (2)
abdominal pain (General disorders) | 4 (5) | 4 (12) | 6 (6)
allergy (General disorders) | 0 (0) | 2 (2) | 0 (0)
anemia (General disorders) | 14 (14) | 13 (13) | 13 (13)
blurred vision (General disorders) | 0 (0) | 0 (0) | 2 (2)
constipation (General disorders) | 1 (1) | 1 (1) | 1 (1)
dehydration (General disorders) | 2 (2) | 0 (0) | 1 (1)
diarrhea (General disorders) | 4 (4) | 5 (6) | 3 (3)
dry mouth (General disorders) | 0 (0) | 2 (2) | 1 (1)
edema (General disorders) | 6 (6) | 3 (3) | 2 (2)
ALT/AST elevated (General disorders) | 8 (13) | 4 (7) | 3 (5)
fever (General disorders) | 5 (6) | 3 (4) | 0 (0)
fluid overload (General disorders) | 1 (1) | 1 (1) | 0 (0)
heme: clot or bleeding (General disorders) | 3 (3) | 3 (4) | 0 (0)
hypotension (General disorders) | 4 (4) | 6 (6) | 5 (6)
irregular menses (General disorders) | 1 (1) | 0 (0) | 0 (0)
kidney/bladder issue (General disorders) | 2 (2) | 3 (3) | 1 (1)
low albumin (General disorders) | 7 (7) | 6 (6) | 6 (6)
metabolic/electrolyte abnormality (General disorders) | 9 (14) | 8 (12) | 9 (13)
MSK pain (General disorders) | 1 (1) | 3 (3) | 0 (0)
Nausea/vomiting (General disorders) | 6 (7) | 3 (3) | 3 (3)
Other GI (General disorders) | 5 (6) | 6 (9) | 3 (3)
other infection (General disorders) | 6 (8) | 5 (8) | 4 (5)
other nervous system (General disorders) | 0 (0) | 0 (0) | 2 (2)
post op pain (General disorders) | 14 (14) | 12 (12) | 11 (11)
psychiatric (General disorders) | 3 (3) | 1 (1) | 3 (3)
respiratory distress (General disorders) | 1 (1) | 3 (3) | 3 (3)
sinus tachycardia (General disorders) | 2 (2) | 2 (2) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-08-08): https://cdn.clinicaltrials.gov/large-docs/97/NCT02713997/Prot_SAP_000.pdf
  • Informed Consent Form (2019-11-25): https://cdn.clinicaltrials.gov/large-docs/97/NCT02713997/ICF_001.pdf